CLINICAL TRIAL: NCT02872662
Title: Individual Molecular Minimal Residual Disease (MRD) Monitoring for Patients With MDS and Mixed MDS/MPN Treated With Allogeneic Stem Cell Transplantation
Brief Title: Individual Molecular MRD Monitoring for MDS Patients After Allo-SCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nordic MDS Group (Network)
Responsible Party: Sponsor
Other Study IDs: NMDSG14B
Record Dates: First submitted 2016-05-02; First posted 2016-08-19 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: MDS; SCT; MRD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to develop highly sensitive methods for early detection of relapse based on the patients unique mutations. Initially, a mutational screen is being performed. Primers directed against these mutations will be constructed and presence of mutations will be followed in bone marrow and blood frequently after transplantation.

DETAILED DESCRIPTION:
This study aims to develop highly sensitive methods for early detection of relapse based on the patients unique mutations.

Screening of mutations In collaboration with Department for clinical genetics, Uppsala, an initial screening of mutations will be performed using the commercial TrueSight© sequencing panel which includes 54 genes recurrently mutated in myeloid diseases. Based on the mutations identified, PCR-primers for all patient-specific mutations will be designed. Patients without any mutation will be excluded from the study. The mutational screen is performed as soon as a patient is being identified as a potential candidate for allogeneic stem cell transplantation (SCT) and evaluated for most optimal pre-SCT treatment. The patient is included in the study before the bone marrow sampling preceding SCT. In case a mutational screen has not been performed before pre-SCT MDS treatment, a mutational screen from the diagnostic national biobank sample (peripheral blood) can be performed.

MRD surveillance After the transplantation, peripheral blood samples will be collected once monthly; and bone marrow samples will be collected at month 1, 3, 6 after SCT followed by sampling every third month until relapse or death. The samples are sent to Biobanking and Molecular Resource Infrastructure of Sweden (bbmri) who will extract DNA and store the samples. By using the highly sensitive digital-PCR method the investigators will determine the size of the different clones at the different time points. In addition to biobanking of DNA, bbmri will collect and vital froze mononuclear cells (MNCs) to be used for experimental studies.

Statistics Landmark analyses will be performed at different time points after SCT, using presence of MRDs as a risk factor included in a multivariate analysis. Furthermore, the investigators will calculate sensitivity, specificity and predictive value for MRDs in relation to relapse. For each specific mutation, with high enough frequency in the cohort, the investigators will define cut-off values of the MRD where relapse is impending.

ELIGIBILITY:
Inclusion Criteria:

1. MDS with allo SCT to be performed
2. One or more mutations identified
3. Written informed consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 consecutive MDS patients undergoing allogeneic SCT
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Level of variant allele frequency (MRD) associated with full hematological relapse | From inclusion up to end of study (August 2019)
  MRD is a quantative variable defined as variant allele frequency of patient-specific mutations. The association between MRD and relapse and survival will be studied.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Hellström-Lindberg, Prof, Principal Investigator — Karolinska Institutet
Locations (8):
- Denmark (2):
  - Department of Hematology, Aarhus University Hospital, Aarhus
  - Department of Hematology, Rigshospitalet Univsersity Hospital, Copenhagen
- Norway (2):
  - Department of Medcine, Haukeland University Hospital, Bergen
  - Department of Hematology, Rikshospitalet University Hospital, Oslo
- Sweden (4):
  - Department of Hematology and Coagulation, Sahlgrenska University hospital, Gothenburg
  - Department of Hematology, Lund University Hospital, Lund
  - Department of Hematology, Karolinska University Hospital, Stockholm
  - Department of Hematology, Akademiska University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Mutational data, MRD and clinical data is planned to be published

REFERENCES:
- [Derived] Tobiasson M, Pandzic T, Illman J, Nilsson L, Westrom S, Ejerblad E, Olesen G, Bjorklund A, Olsnes Kittang A, Werlenius O, Lorentz F, Rasmussen B, Cammenga J, Weber D, Lindholm C, Wiggh J, Dimitriou M, Moen AE, Yip Lundstrom L, von Bahr L, Baltzer-Sollander K, Jadersten M, Kytola S, Walldin G, Ljungman P, Groenbaek K, Mielke S, Jacobsen SEW, Ebeling F, Cavelier L, Smidstrup Friis L, Dybedal I, Hellstrom-Lindberg E. Patient-Specific Measurable Residual Disease Markers Predict Outcome in Patients With Myelodysplastic Syndrome and Related Diseases After Hematopoietic Stem-Cell Transplantation. J Clin Oncol. 2024 Apr 20;42(12):1378-1390. doi: 10.1200/JCO.23.01159. Epub 2024 Jan 17. PMID 38232336